CLINICAL TRIAL: NCT04896476
Title: Prospective Feasibility Study Evaluating EchoMark LP Placement and EchoSure Measurements for Subjects Requiring Arteriovenous Fistulae
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sonavex, Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDE-F1-2021; R44HL147423 (NIH)
Record Dates: First submitted 2021-05-10; First posted 2021-05-21 (Actual); Results first posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-12

CONDITIONS: Kidney Diseases; Arteriovenous Fistula
MeSH Terms: conditions — Kidney Diseases; Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- EchoMark/EchoSure (Experimental): All subjects will undergo a physician exam prior an arteriovenous fistula creation per the institution's standard of care. After the fistula creation is completed, but prior to closure, the EchoMark will be implanted under the outflow vein.
  The follow-up EchoSure scans will be conducted by the designated EchoSure user without the investigator and without the sonographer/RVT conducting the Duplex exam in the room, either during the routine work-up prior to the surgeon seeing the patient or after. The EchoSure results for flow, and vessel depth and diameter are shown as numerical values on the screen of the EchoSure device.
  Interventions: Device: EchoMark / EchoSure

INTERVENTIONS:
Device: EchoMark / EchoSure — The EchoMark is to be secured a minimum of 3 cm away from the anastomosis.
  The follow-up EchoSure scans will be conducted by the designated EchoSure user without the investigator and without the sonographer/RVT conducting the Duplex exam in the room, either during the routine work-up prior to the surgeon seeing the patient or after. The EchoSure results for flow, and vessel depth and diameter are shown as numerical values on the screen of the EchoSure device.

SUMMARY:
Multi-center trial to assess the feasibility and safety of the EchoMark LP and the EchoMark diagnostic ultrasound system for assessing AV fistula blood flow, diameter, and depth.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm, non-blinded clinical trial designed to evaluate the feasibility and safety of the EchoMark and the EchoSure in subjects undergoing new upper arm autologous arteriovenous fistula creation who require hemodialysis. All subjects will provide informed consent prior to undergoing any study procedures. The study will consists of multiple follow-up visits during the 52 week duration. Subjects are able to re-consent and remain in follow-up for an additional year.

ELIGIBILITY:
Inclusion Criteria:

1. Males or non-pregnant, non-breastfeeding females ≥ 18 years of age but < 85 years of age at the time of informed consent
2. Subject is able and willing to provide written informed consent prior to receiving any non-standard of care, protocol specific procedures
3. Subject is willing and capable of complying with all required follow-up visits
4. Subject and/or Care Team agree that the distance and transportation resources from the subject's home to the clinic are reasonable for study participation and compliance
5. Subject has an estimated life expectancy > 18 months
6. Subject is ambulatory (cane or walker are acceptable)
7. Subjects presenting for upper arm autologous arteriovenous fistula creation
8. Vein diameter > 2.5 mm at the antecubital fossa via imaging
9. Artery diameter > 3 mm via imaging
10. Subject is not participating in another investigational clinical trial that has not met its primary endpoint. Participation in a post-market registry is acceptable.

Exclusion Criteria:

1. Subjects receiving a forearm fistula.
2. Subject has history of Steal Syndrome.
3. Subject who is immunocompromised or immunosuppressed.
4. Subject has had three previous failed AV fistulae for hemodialysis access
5. Subjects expecting to undergo major surgery within 60 days from the EchoMark implantation.
6. Known or suspected active infection on the day of the index procedure.
7. Subjects who had infection(s) in the 30-day window prior to EchoMark placement to reduce the likelihood of partially treated infections that can seed the device and fistula
8. Subjects with diagnosed bleeding disorder, thrombocytopenia (platelet count <50,000), hypercoagulability, and history of recurrent deep vein thrombosis not related to AV access
9. Subjects with active malignancy
10. Subjects with a history of poor compliance with the dialysis protocol
11. Subjects with a known or suspected allergy to any of the device materials
12. Subjects with an existing fistula or graft
13. Subjects who are pregnant, plan to become pregnant, or are breastfeeding.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2025-06-06 (Estimated)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Trinity Research Group, Dothan, Alabama
  - SKI Vascular Center, Peoria, Arizona
  - Michgan Vascular Center, Flint, Michigan
  - Surgical Specialist of Charlotte, Charlotte, North Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- EchoMark: All subjects will undergo a physician exam prior an arteriovenous fistula creation per the institution's standard of care. After the fistula creation is completed, but prior to closure, the EchoMark will be implanted under the outflow vein.
  EchoMark: The EchoMark is to be secured a minimum of 3 cm away from the anastomosis.
Period: Overall Study
Arm/Group | EchoMark
Started | 20
Completed | 17
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | EchoMark
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 64.3 [40 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 11
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint
Description: Composite of new major device related adverse events (MAEs) at 30 days post EchoMark implantation, as adjudicated by the Clinical Events Committee (CEC) including:
  * Device or procedure-related death
  * Device related infection
  * Device related interventions
  * Device related hospitalizations
  * Fistula failure
  * Fistula rupture
  * Aneurysm
Time Frame: 30 Days
Measure: Number; unit: MAES within 30 days post baseline visit
Arm/Group | EchoMark
Number analyzed (Participants) | 20
MAES within 30 days post baseline visit | 0

2. Primary Outcome: Primary Feasibility Endpoint
Description: Rate of Technical Success defined as the successful implantation of the EchoMark implant. Technical success will be assessed from baseline to 4 months.
Time Frame: 4 Months
Measure: Count of Participants; unit: Participants
Arm/Group | EchoMark
Number analyzed (Participants) | 20
Participants | 20

3. Primary Outcome: Rate of Technical Success Defined as the Successful Ability to Determine Blood Flow, Diameter, and Depth Measurements Using the EchoSure Diagnostic Ultrasound System. Technical Success Will be Assessed From Baseline to 4 Months.
Description: Rate of Technical Success defined as the successful ability to determine blood flow, diameter, and depth measurements using the EchoSure diagnostic ultrasound system. Technical success will be assessed from baseline to 4 months.
Time Frame: 4 Months
Measure: Count of Units; unit: EchoSure Scans
Units Other Than Participants: EchoSure Scans
Groups:
- EchoMark: All subjects will undergo a physician exam prior an arteriovenous fistula creation per the institution's standard of care. After the fistula creation is completed, but prior to closure, the EchoMark will be implanted under the outflow vein.
  The follow-up EchoSure scans will be conducted by the designated EchoSure user without the investigator and without the sonographer/RVT conducting the Duplex exam in the room, either during the routine work-up prior to the surgeon seeing the patient or after. The EchoSure results for flow, and vessel depth and diameter are shown as numerical values on the screen of the EchoSure device.
Arm/Group | EchoMark
Number analyzed (Participants) | 20
Number analyzed (EchoSure Scans) | 273
EchoSure Scans | 270

4. Other Pre Specified Outcome: Comparison of EchoSure and Duplex Measurements Using Percentages
Description: Bland Altman using percentages will assess the agreement between two measurements.
  Only duplex images that pass the CoreLab quality control check will be included in the assessment.
  The results will be calculated as a percent difference between the two measurements with a value of zero corresponding to exact agreement.
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: Flow Rate Percent Difference
Arm/Group | EchoMark
Number analyzed (Participants) | 20
Flow Rate Percent Difference | -7.8 (38.5)

5. Other Pre Specified Outcome: Comparison of EchoSure and Duplex Measurements of Diameter
Description: as for outcome 4
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: Diameter Percent Difference
Arm/Group | EchoMark
Number analyzed (Participants) | 20
Diameter Percent Difference | 9.4 (19.7)

6. Other Pre Specified Outcome: Comparison of EchoSure and Duplex Measurements of Depth
Description: as for outcome 4
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: Depth Percent Difference
Arm/Group | EchoMark
Number analyzed (Participants) | 20
Depth Percent Difference | 18.4 (23.8)

7. Other Pre Specified Outcome: Comparison of EchoSure Depth Measurements to Independent Reviewer Measured Depth Results.
Description: Bland Altman using percentages will assess the agreement between two measurements.
  The results will be calculated as a percent difference between the two measurements with a value of zero corresponding to exact agreement.
Time Frame: 4 Months
Measure: Mean (Standard Deviation); unit: Depth Percent Difference
Arm/Group | EchoMark
Number analyzed (Participants) | 20
Depth Percent Difference | 18.4 (23.8)

8. Other Pre Specified Outcome: Time to Radiographic Maturation
Description: defined as the number of days from baseline procedure to date of radiographic maturation (date of ultrasound imaging, as adjudicated by the CEC). Radiographic maturation is defined as a fistula with volume flow of 500mL/min and 5mm diameter.
Time Frame: 12 Months
Population: One subject never reached clinical maturation
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | EchoMark
Number analyzed (Participants) | 19
Number of Days | 28.8 (23.4)

9. Other Pre Specified Outcome: Time to Clinical Maturation
Description: defined as the number of days from baseline procedure to date of clinical maturation. Clinical maturation is defined as 75% of dialysis sessions with successful 2 needle cannulation. Date of clinical maturation is defined as first date of the 4-week window when clinical maturation is achieved.
Time Frame: 12 Months
Population: Analysis included subjects with supporting cannulation records
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | EchoMark
Number analyzed (Participants) | 7
Number of Days | 67.5 (4.9)

10. Other Pre Specified Outcome: Radiographic Maturation Success Rate
Description: defined as the percentage of subjects that achieve radiographic maturation (as determined by the physician and adjudicated by the CEC) by end of study. Radiographic maturation is defined as a fistula with 500mL/min and 5mm diameter.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | EchoMark
Number analyzed (Participants) | 20
Participants | 19

11. Other Pre Specified Outcome: Clinical Maturation Success Rate
Description: defined as the percentage of subjects that achieve clinical maturation by end of study. Date of clinical maturation is defined as first date of the 4-week window when clinical maturation is achieved.
Time Frame: 12 Months
Population: 17 subjects were cleared for cannulation and source documents were requested. 2 subjects did not require dialysis treatment. Records were obtained for 7 Subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | EchoMark
Number analyzed (Participants) | 7
Participants | 7

12. Other Pre Specified Outcome: Number of Patients With 6-Month Patency
Description: defined by the status (yes/no) of an arteriovenous dialysis access with detectable blood flow through and beyond the anastomosis shown by either an imaging modality or physical examination (presence of a palpable thrill or audible bruit along some point of the arteriovenous dialysis access beyond the arteriovenous anastomosis).
Time Frame: 6 Months
Population: Subjects who completed the 6-month visit.
Measure: Count of Participants; unit: Participants
Arm/Group | EchoMark
Number analyzed (Participants) | 16
Participants | 16

13. Other Pre Specified Outcome: Number of Patients With 12-Month Patency
Description: as for outcome 12
Time Frame: 12 Months
Population: Subjects who completed the 12-month visit
Measure: Count of Participants; unit: Participants
Arm/Group | EchoMark
Number analyzed (Participants) | 16
Participants | 16

14. Other Pre Specified Outcome: Occurrence of Events Occurring Within 30 Days of Implantation That Require Reinterventions (Open or Endovascular), Hospitalizations, or Prolongation of Existing Hospitalization.
Time Frame: 30 Days
Measure: Number; unit: Events
Arm/Group | EchoMark
Number analyzed (Participants) | 20
Events | 1

15. Other Pre Specified Outcome: Occurrence of Events of Reported Reduction of Blood Flow That Prevents the Ability to Cannulate or Requires Further Assessment and/or Intervention From Baseline Procedure to 12 Months.
Time Frame: 12 Months
Measure: Number; unit: Events
Arm/Group | EchoMark
Number analyzed (Participants) | 20
Events | 4

16. Other Pre Specified Outcome: Occurrence of the Reported Inability to Cannulate Fistula Beginning Once the Fistula is Deemed Radiographically and Clinically Mature to 12 Months.
Time Frame: 12 Months
Population: Subjects that have been deemed clinically mature
Measure: Number; unit: Occurrence of Event
Arm/Group | EchoMark
Number analyzed (Participants) | 7
Occurrence of Event | 0

17. Other Pre Specified Outcome: Occurrence of Events of the Development of Steal Syndrome From Baseline to 12 Months.
Time Frame: 12 Months
Measure: Number; unit: Events
Arm/Group | EchoMark
Number analyzed (Participants) | 20
Events | 1

18. Other Pre Specified Outcome: Occurrence of Events of Bleeding Requiring Surgical Intervention (Including PRBC Transfusion) From Baseline to 12 Months.
Time Frame: 12 Months
Measure: Number; unit: Events
Arm/Group | EchoMark
Number analyzed (Participants) | 20
Events | 0

19. Other Pre Specified Outcome: Occurrence of Events of Infiltration Requiring Procedural Intervention From Baseline to 12 Months.
Time Frame: 12 Months
Measure: Number; unit: Events
Arm/Group | EchoMark
Number analyzed (Participants) | 20
Events | 2

20. Other Pre Specified Outcome: Occurrence of Events of Hematoma Requiring Procedural Intervention From Baseline to 12 Months.
Time Frame: 12 Months
Measure: Number; unit: Events
Arm/Group | EchoMark
Number analyzed (Participants) | 20
Events | 0

21. Other Pre Specified Outcome: Occurrence of Events of the Inability to Use the EchoSure Component of the System From Baseline to 4 Months
Description: Due to:
  1. Migration of the EchoMark device
  2. Early resorption of the EchoMark device as defined as breakdown of the EchoMark shape prior to 4 months from index procedure.
Time Frame: 4 Months
Measure: Number; unit: Events
Arm/Group | EchoMark
Number analyzed (Participants) | 20
Events | 0

22. Other Pre Specified Outcome: Occurrence of Events of Pain Related to the Study Devices From Baseline to 12 Months
Time Frame: 12 Months
Measure: Number; unit: Events
Arm/Group | EchoMark
Number analyzed (Participants) | 20
Events | 1

23. Other Pre Specified Outcome: Occurrence of Events of Infection (Not Limited to Infection Requiring Implant Explanation) From Baseline to 12 Months
Time Frame: 12 Months
Measure: Number; unit: Events
Arm/Group | EchoMark
Number analyzed (Participants) | 20
Events | 0

24. Other Pre Specified Outcome: Occurrence of Events of Infection Confirmed by Either Implant Explanation or Purulent Fluid on Pathologic Assessment During Incision and Drainage Beginning at Baseline to 12 Months
Time Frame: 12 Months
Measure: Number; unit: Events
Arm/Group | EchoMark
Number analyzed (Participants) | 20
Events | 0

25. Other Pre Specified Outcome: Composite of New Major Device Related Adverse Events (MAEs) at 12 Months Post EchoMark LP Implantation, as Adjudicated by the Clinical Events Committee (CEC).
Description: The proportion of subjects with device success and free from device- and/or procedure related
  SAEs (per CEC adjudication) at 12 months including:
  * Device or procedure-related death
  * Device related infection
  * Device related interventions
  * Device related hospitalizations
  * Fistula failure
  * Fistula rupture
  * Aneurysm
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | EchoMark
Number analyzed (Participants) | 20
Participants | 15

ADVERSE EVENTS:
Time Frame: The study duration was originally for 1 year. Adverse Events for all 20 subjects were reported for 1 year. Subjects were able to re-consent for an additional year of follow-up and adverse events were/ are being reported for an additional year for all subjects who re-consented.
Description: All adverse events were assessed by the site primary investigator and adjudicated by the CEC.
Arm/Group | EchoMark
All-Cause Mortality (participants affected / at risk) | 3/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 16/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EchoMark (N=20)
Seroma (Surgical and medical procedures) | 0 (0)
Fluid Collection (Vascular disorders) | 2 (2)
Stenosis (Vascular disorders) | 12 (24)
Pain (including cannulation-related pain) (Surgical and medical procedures) | 4 (4)
Restenosis (Vascular disorders) | 3 (5)
Reduction in Blood Flow (Vascular disorders) | 4 (4)
Numbness, Tingling (Surgical and medical procedures) | 1 (1)
Steal Syndrome (Vascular disorders) | 1 (1)
Infiltration (Injury, poisoning and procedural complications) | 5 (5)
Difficulty Cannulating (Injury, poisoning and procedural complications) | 4 (4)
Malfunctioning Catheter (Vascular disorders) | 1 (1)
Excessive Bleeding (Vascular disorders) | 1 (1)
In-Stent Restenosis (Vascular disorders) | 1 (1)
Poor Maturation (Vascular disorders) | 1 (1)
Swelling Access Extremity (Vascular disorders) | 1 (1)
Inability to Cannulate (Vascular disorders) | 1 (1)
Blockage Left Leg (Vascular disorders) | 1 (1)
Fluid Overload (Vascular disorders) | 2 (2)
Non-Maturing Fistula (Vascular disorders) | 1 (1)
Back Pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT04896476/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT04896476/ICF_001.pdf